CLINICAL TRIAL: NCT03260647
Title: Risk Stratified Multidisciplinary Ambulatory Management of Malignant Bowel Obstruction (MAMBO) Program for Women With Advanced Gynecological Cancers
Brief Title: Risk Stratified Multidisciplinary Ambulatory Management of Malignant Bowel Obstruction in Gynecological Cancers
Acronym: MAMBO
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: MAMBO
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients with MBO who undergo palliative procedures or surgical intervention will be offered optional consent for tissue collection for research. Fresh-frozen and formalin-fixed paraffin-embedded (FFPE) tumour tissue specimens, as well as ascites will be collected for translational studies. Stool samples will be collected for microbiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Management algorithm for Malignant Bowel Obstruction — a proposed management algorithm for MBO has been developed to provide a pathway that safeguards quality and continuity of care for patients under a multidisciplinary team. It will engage key-stakeholders and foster an inter-professional approach. It incorporates an in-patient management algorithm and a novel nursing-led ambulatory management algorithm to supplement patient's medical management

SUMMARY:
Management of Malignant Bowel Obstruction (MBO) in Patients with Advanced Gynecological Cancers

DETAILED DESCRIPTION:
Guidelines for the management of patients with Malignant Bowel Obstruction(MBO) are not available and as such, there remains an urgent need for a collaborative approach to streamline patient care and optimize use of hospital resources. This study will focus on management of MBO in advanced gynecological cancers.If patients with MBO can be effectively managed in an ambulatory setting, this may improve quality and consistency of patient care, and help reduce volume and duration of bed occupancy.

ELIGIBILITY:
Inclusion Criteria:

Histologically and /or cytologically confirmed gynecological cancer, including ovarian, fallopian tube, endometrial, cervical or primary peritoneal cancer Deemed to be at risk of developing or have a clinical diagnosis of MBO as defined using the following criteria: clinical evidence of bowel obstruction (history/physical/radiological examination; and bowel obstruction beyond the ligament of Treitz.

Exclusion Criteria:

There are no specified exclusion criteria for this study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with gynecological cancer and at risk or presently having Malignant bowel obstruction (MBO)
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Optimization of multidisciplinary care | 2 years
  To optimize the multidisciplinary care management of MBO in patients with advanced gynecological cancer treated at University Health Network (UHN) which include in-patient and ambulatory management algorithm for MBO
  • Measured by a ratio of days alive and out of hospital compare to days in hospital within the first 60 days after diagnosis of MBO

SECONDARY OUTCOMES:
Evaluation of treatment outcomes | 2 years
  To evaluate the treatment outcomes of patients with MBO
  * Measured by resolution of MBO and overall survival
  * Measured by transition through specific bowel management colour code system
Evaluation of impact of MBO management on hospital visits | 2 years
  To evaluate the impact of MBO management on number of emergency room visits, hospital admission and number of days alive and outside of hospital within the first 168 days (6 months) after the diagnosis of MBO
Evaluation of impact of MBO management on patient reported outcomes | 2 years
  To evaluate the impact of ambulatory MBO management on patient reported outcomes using the Distress Assessment & Response Tool (DART)
To evaluate nutritional status of patients with MBO | 2 years
  To evaluate the nutritional status of patients with MBO
  • Measured by monthly albumin and weight
Evaluation of clinico-pathological factors | 2 years
  To evaluate the clinico-pathological factors that may predict benefit from palliative surgery, chemotherapy and total parenteral nutrition (TPN)
Improve patient understanding and awareness of MBO | 2 years
  To improve patients' understanding and awareness of MBO with patient education material.
Determine percentage number of patient microbiome sample analyses completed | 1.5 years
  To record the percentage of patients who agree to, and for whom sample collection and analysis is completed
Record changes in the sum and types of gut microbiome from baseline to study end | 1.5 years
  Changes in the sum as well as types of microbiomes as recorded at baseline, initiation of total parenteral nutrition, incidence of an MBO and end of study are to be recorded
Evaluate cannabis use in patient population | 1.5 years
  Assess for any relationship between cannabis use and MBO

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran E, Spiceland C, Sandhu NP, Jatoi A. Malignant Bowel Obstruction in Patients With Recurrent Ovarian Cancer. Am J Hosp Palliat Care. 2016 Apr;33(3):272-5. doi: 10.1177/1049909114566225. Epub 2014 Dec 31. PMID 25552305
- [Background] Mooney SJ, Winner M, Hershman DL, Wright JD, Feingold DL, Allendorf JD, Neugut AI. Bowel obstruction in elderly ovarian cancer patients: a population-based study. Gynecol Oncol. 2013 Apr;129(1):107-12. doi: 10.1016/j.ygyno.2012.12.028. Epub 2012 Dec 26. PMID 23274561
- [Background] Sartori E, Chiudinelli F, Pasinetti B, Maggino T. Bowel obstruction and survival in patients with advanced ovarian cancer: analysis of prognostic variables. Int J Gynecol Cancer. 2009 Jan;19(1):54-7. doi: 10.1111/IGC.0b013e318198ff4b. No abstract available. PMID 19258942
- [Background] Jayson GC, Kohn EC, Kitchener HC, Ledermann JA. Ovarian cancer. Lancet. 2014 Oct 11;384(9951):1376-88. doi: 10.1016/S0140-6736(13)62146-7. Epub 2014 Apr 21. PMID 24767708
- [Background] Martin-Lorente C, Mackay H, Lafromboise L, et al: Retrospective review of malignant bowel obstruction (MBO) outcomes in patients with epithelial ovarian carcinoma (EOC), International Journal of Gynecological Cancer, 2015, pp 1434-1435
- [Background] Anthony T, Baron T, Mercadante S, Green S, Chi D, Cunningham J, Herbst A, Smart E, Krouse RS. Report of the clinical protocol committee: development of randomized trials for malignant bowel obstruction. J Pain Symptom Manage. 2007 Jul;34(1 Suppl):S49-59. doi: 10.1016/j.jpainsymman.2007.04.011. Epub 2007 Jun 4. PMID 17544243
- [Background] Ripamonti C, Twycross R, Baines M, Bozzetti F, Capri S, De Conno F, Gemlo B, Hunt TM, Krebs HB, Mercadante S, Schaerer R, Wilkinson P; Working Group of the European Association for Palliative Care. Clinical-practice recommendations for the management of bowel obstruction in patients with end-stage cancer. Support Care Cancer. 2001 Jun;9(4):223-33. doi: 10.1007/s005200000198. PMID 11430417
- [Background] Tuca A, Guell E, Martinez-Losada E, Codorniu N. Malignant bowel obstruction in advanced cancer patients: epidemiology, management, and factors influencing spontaneous resolution. Cancer Manag Res. 2012;4:159-69. doi: 10.2147/CMAR.S29297. Epub 2012 Jun 13. PMID 22904637
- [Background] Daniele A, Ferrero A, Fuso L, Mineccia M, Porcellana V, Vassallo D, Biglia N, Menato G. Palliative care in patients with ovarian cancer and bowel obstruction. Support Care Cancer. 2015 Nov;23(11):3157-63. doi: 10.1007/s00520-015-2694-9. Epub 2015 Mar 25. PMID 25805450
- [Background] Ripamonti CI, Easson AM, Gerdes H. Management of malignant bowel obstruction. Eur J Cancer. 2008 May;44(8):1105-15. doi: 10.1016/j.ejca.2008.02.028. Epub 2008 Mar 21. PMID 18359221
- [Background] Cousins SE, Tempest E, Feuer DJ. Surgery for the resolution of symptoms in malignant bowel obstruction in advanced gynaecological and gastrointestinal cancer. Cochrane Database Syst Rev. 2016 Jan 4;2016(1):CD002764. doi: 10.1002/14651858.CD002764.pub2. PMID 26727399
- [Background] Feuer DJ, Broadley KE, Shepherd JH, Barton DP. Surgery for the resolution of symptoms in malignant bowel obstruction in advanced gynaecological and gastrointestinal cancer. Cochrane Database Syst Rev. 2000;(4):CD002764. doi: 10.1002/14651858.CD002764. PMID 11034757
- [Background] Furnes B, Svensen R, Helland H, Ovrebo K. Challenges and outcome of surgery for bowel obstruction in women with gynaecologic cancer. Int J Surg. 2016 Mar;27:158-164. doi: 10.1016/j.ijsu.2016.02.002. Epub 2016 Feb 4. PMID 26853847
- [Background] Levy M, Smith T, Alvarez-Perez A, Back A, Baker JN, Beck AC, Block S, Dalal S, Dans M, Fitch TR, Kapo J, Kutner JS, Kvale E, Misra S, Mitchell W, Portman DG, Sauer TM, Spiegel D, Sutton L, Szmuilowicz E, Taylor RM, Temel J, Tickoo R, Urba SG, Weinstein E, Zachariah F, Bergman MA, Scavone JL. Palliative Care Version 1.2016. J Natl Compr Canc Netw. 2016 Jan;14(1):82-113. doi: 10.6004/jnccn.2016.0009. PMID 26733557
- [Background] Kolomainen DF, Daponte A, Barton DP, Pennert K, Ind TE, Bridges JE, Shepherd JH, Gore ME, Kaye SB, Riley J. Outcomes of surgical management of bowel obstruction in relapsed epithelial ovarian cancer (EOC). Gynecol Oncol. 2012 Apr;125(1):31-6. doi: 10.1016/j.ygyno.2011.11.007. Epub 2011 Nov 12. PMID 22082991
- [Background] Mangili G, Aletti G, Frigerio L, Franchi M, Panacci N, Vigano R, DE Marzi P, Zanetto F, Ferrari A. Palliative care for intestinal obstruction in recurrent ovarian cancer: a multivariate analysis. Int J Gynecol Cancer. 2005 Sep-Oct;15(5):830-5. doi: 10.1111/j.1525-1438.2005.00144.x. PMID 16174232
- [Background] Goto T, Takano M, Aoyama T, Miyamoto M, Watanabe A, Kato M, Sasaki N, Hirata J, Sasa H, Furuya K. Outcomes of palliative bowel surgery for malignant bowel obstruction in patients with gynecological malignancy. Oncol Lett. 2012 Nov;4(5):883-888. doi: 10.3892/ol.2012.835. Epub 2012 Jul 30. PMID 23162616
- [Background] Kucukmetin A, Naik R, Galaal K, Bryant A, Dickinson HO. Palliative surgery versus medical management for bowel obstruction in ovarian cancer. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD007792. doi: 10.1002/14651858.CD007792.pub2. PMID 20614464
- [Background] Bryan DN, Radbod R, Berek JS. An analysis of surgical versus chemotherapeutic intervention for the management of intestinal obstruction in advanced ovarian cancer. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):125-34. doi: 10.1111/j.1525-1438.2006.00283.x. PMID 16445622
- [Background] Diver E, O'Connor O, Garrett L, Boruta D, Goodman A, Del Carmen M, Schorge J, Mueller P, Growdon W. Modest benefit of total parenteral nutrition and chemotherapy after venting gastrostomy tube placement. Gynecol Oncol. 2013 May;129(2):332-5. doi: 10.1016/j.ygyno.2013.02.002. Epub 2013 Feb 8. PMID 23402902
- [Background] Chouhan J, Gupta R, Ensor J, Raghav K, Fogelman D, Wolff RA, Fisch M, Overman MJ. Retrospective analysis of systemic chemotherapy and total parenteral nutrition for the treatment of malignant small bowel obstruction. Cancer Med. 2016 Feb;5(2):239-47. doi: 10.1002/cam4.587. Epub 2015 Dec 29. PMID 26714799
- [Background] Abu-Rustum NR, Barakat RR, Venkatraman E, Spriggs D. Chemotherapy and total parenteral nutrition for advanced ovarian cancer with bowel obstruction. Gynecol Oncol. 1997 Mar;64(3):493-5. doi: 10.1006/gyno.1996.4605. PMID 9062158
- [Background] Li M, Macedo A, Crawford S, Bagha S, Leung YW, Zimmermann C, Fitzgerald B, Wyatt M, Stuart-McEwan T, Rodin G. Easier Said Than Done: Keys to Successful Implementation of the Distress Assessment and Response Tool (DART) Program. J Oncol Pract. 2016 May;12(5):e513-26. doi: 10.1200/JOP.2015.010066. Epub 2016 Apr 5. PMID 27048610
- [Background] Brard L, Weitzen S, Strubel-Lagan SL, Swamy N, Gordinier ME, Moore RG, Granai CO. The effect of total parenteral nutrition on the survival of terminally ill ovarian cancer patients. Gynecol Oncol. 2006 Oct;103(1):176-80. doi: 10.1016/j.ygyno.2006.02.013. Epub 2006 Mar 27. PMID 16564074
- [Derived] Madariaga A, Jivraj N, Soberanis Pina P, Somji F, Truong T, Melwani S, Lovas M, Gogos TA, Sajewycz K, Bhat G, Alqaisi H, Gonzalez-Ochoa E, Veneziani A, Garg V, Dhani NC, Grant R, Bowering V, Oza AM, Wang L, Berlin A, Lheureux S. Electronic malignant bowel obstruction symptom monitoring smartphone application for patients with gynecologic cancers. Int J Gynecol Cancer. 2024 Oct 7;34(10):1612-1618. doi: 10.1136/ijgc-2024-005490. PMID 38821545
- [Derived] Cusimano MC, Sajewycz K, Nelson M, Jivraj N, Lee YC, Bowering V, Oza A, Lheureux S, Ferguson SE. Supported self-management as a model for end-of-life care in the setting of malignant bowel obstruction: A qualitative study. Gynecol Oncol. 2020 Jun;157(3):745-753. doi: 10.1016/j.ygyno.2020.03.009. Epub 2020 Mar 23. PMID 32217004